CLINICAL TRIAL: NCT06022198
Title: Study of Bronchoalveolar Lavage in Patients Recovered From COVID-19 Pneumonia
Brief Title: Bronchoalveolar Lavage in Recovered From COVID-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Abd Elmoniem Mohamed (Other)
Collaborators: Marwa Salah Abdelrazek Ghanem (Unknown); Mohammad Khairy El-Badrawy (Unknown); Tamer Ali Elhadidy (Unknown); Dalia Abdellateif Abdelghany (Unknown)
Responsible Party: Sponsor-Investigator, Mohamed Abd Elmoniem Mohamed, Assistant lecturer, Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD.21.01.408
Record Dates: First submitted 2023-08-31; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Bronchoalveolar Lavage
Keywords: Bronchoalveolar lavage; COVID-19 Pneumonia
MeSH Terms: interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Intervention Model Description: prospective cross sectional study at which COVID-19 patients with persistent pulmonary infiltrate one month after discharge from isolation department at Mansoura university hospitals will be enrolled in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recovered From COVID-19 Pneumonia (Experimental): Bronchoalveolar Lavage in Recovered From COVID-19 Pneumonia
  Interventions: Procedure: Bronchoalveolar Lavage

INTERVENTIONS:
Procedure: Bronchoalveolar Lavage — Bronchoalveolar Lavage

SUMMARY:
Coronaviruses such as SARS-CoV2, MERS-CoV, and SARS-CoV can cause significant morbidity and mortality in infected persons. Lung is the most common site of infection for these viruses, which may manifest as acute respiratory distress syndrome and mortality. Pulmonary involvement is also responsible for the high viral transmission The aim of this study is to evaluate BAL in post-acute COVID-19 patients for:Cytological and cellular patterns. Microbial analysis for possibility of presence of bacterial, mycobacerial or fungal co-infection.PCR for corona virus

DETAILED DESCRIPTION:
On December 31, 2019, a cluster of cases of pneumonia in people who were later linked to Wuhan Seafood Market in Wuhan, Hubei, China, were reported. Just a week later, Chinese health authorities confirmed that those cases were caused by a novel coronavirus, later named as SARS-CoV2 .

Till date, six coronavirus species are known to cause human diseases. Four of the already-known coronavirus species, i.e., 229E, OC43, NL63, and HKU1, are commonly circulating viruses in human population and cause mild common cold-like symptoms.

Two of the already-known strains of coronavirus, severe acute respiratory syndrome-coronavirus (SARS-CoV) and Middle East respiratory syndrome-CoV (MERS-CoV) are zoonotic in origin and cause serious illnesses which can be fatal.

Coronaviruses such as SARS-CoV2, MERS-CoV, and SARS-CoV can cause significant morbidity and mortality in infected persons. Lung is the most common site of infection for these viruses, which may manifest as acute respiratory distress syndrome and mortality. Pulmonary involvement is also responsible for the high viral transmission.

BAL, bronchial wash, and protected specimen brush are bronchoscopic procedures used to provide microbiological samples from lower respiratory airways. However, because of the risk of viral transmission, bronchoscopy is not routinely indicated for the diagnosis of COVID-19.

Even if SARS-CoV-2 shares similarities with the other coronaviruses, the higher diffusion rate and the possibility to induce fatal complications, such as severe pneumonia, acute respiratory distress syndrome (ARDS), thrombosis, septic shock and organ failure, make this virus a major public health threat.

Since the first guidelines for autopsy on both confirmed and suspected COVID-19-positive patients were published in February 2020, an increasing number of biopsies and autopsies have been performed. However, our knowledge regarding the precise nature of the immunological defense in various organ systems in response to viral infection, as well as the response patterns in specific tissues, is largely incomplete but is essential in order to initiate timely and targeted antiviral, anti-inflammatory, anticoagulative, or even antifibrotic therapy .

As of yet, most research papers have focused on the inflammatory status at the plasma level of COVID-19 patients. However, because the main target organ is the lung, it is crucial to understand the inflammatory status at the deep lung level during different stages of the infection. Currently, limited data are available about alveolar inflammatory status in COVID-19 patients because of concerns in relation to using bronchoscopy to avoid aerosol generation. The aim of this study is to evaluate BAL in post-acute COVID-19 patients for:Cytological and cellular patterns. Microbial analysis for possibility of presence of bacterial, mycobacerial or fungal co-infection.PCR for corona virus

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent pulmonary infiltrate one month after discharge from isolation building at Mansoura university hospitals, previously tested positive for SARS-CoV-2 infection by real-time PCR on nasopharyngeal swab during admission, discharged and discontinued transmission based precautions according to CDC guidance:

Symptom-Based Strategy for Discontinuing Transmission-Based Precautions (CDC, 2020)

Patients with mild to moderate illness who are not severely immunocompromised:

* At least 10 days have passed since symptoms first appeared and
* At least 24 hours have passed since last fever without the use of fever-reducing medications and
* Symptoms (e.g., cough, shortness of breath) have improved

Patients with severe to critical illness or who are severely immunocompromised1:

* At least 10 days and up to 20 days have passed since symptoms first appeared and
* At least 24 hours have passed since last fever without the use of fever-reducing medications and
* Symptoms (e.g., cough, shortness of breath) have improved
* Consider consultation with infection control experts

Exclusion Criteria:

* Age: patients less than 18 years old.
* Patient refuse to undergo bronchoscopy.
* Patients unfit for bronchoscopy (hemodynamic instability, recent myocardial infarction, severe hypoxia, uncooperative patient, severe bleeding disorder).
* Patients known to have chronic airway pulmonary diseases or interstitial lung diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
evaluate BAL in post-acute COVID-19 patients | Baseline
  Understanding the pathophysiological mechanisms of COVID-19 and nature of the immunological defense in lungs in response to viral infection by SARS-CoV2 is essential in order to initiate timely and targeted anti-inflammatory, anticoagulative, or even antifibrotic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ghanem, Principal Investigator — Mansoura university Faculty of medicine
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No